CLINICAL TRIAL: NCT02192112
Title: Evaluation of Transcutaneous Stimulation of Lumbosacral Nerve Roots: A Pilot Study
Brief Title: Advanced XLIF Monitoring Pilot Study
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.NV1301
Record Dates: First submitted 2014-07-01; First posted 2014-07-16 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Lumbar Disc Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Though the utility of NVM5 neuromonitoring by stimulating within the surgical site during XLIF has been demonstrated, it is hypothesized that more information may be gathered if a greater section of the motor neural pathway was monitored (i.e., stimulation above the surgical site and recording the subsequent muscle response in the lower limbs). Currently, there has not been demonstrated a practical method of stimulating the lumbosacral nerve roots locally, but well-above the surgical site in this fashion.

This protocol is intended to evaluate the feasibility and reproducibility of using surface stimulation and return (anode) electrodes to stimulate the lumbosacral nerve roots, and record responses from the relevant innervated muscle groups of the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female spine surgery patients who are at least 18 years of age
2. Surgical candidates for lateral approach lumbar spine surgery at spinal levels L2 to L5, inclusive of L4-5
3. Patients who understand the conditions of enrollment and are willing to sign an informed consent to participate in the evaluation

Exclusion Criteria:

1. Currently undergoing surgical treatment at any spinal level other than L2 to L5, including S1
2. Pregnant women
3. Implanted pacemaker, defibrillator, or other electronic devices
4. Involved in active litigation relating to the spine (worker's compensation claim is allowed if it is not contested)
5. Underlying neurological disease or neurological deficit that is not associated with the condition for which he/she is seeking surgical intervention (e.g., diabetic peripheral neuropathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 20 subjects will be consecutively enrolled in this prospective pilot study from up to three (3) participating centers. Patients who, in the surgeon investigator's opinion, require lateral approach spinal fusion surgery at spinal level L4-5 (though may include any number of levels from L2 through L5), and have consented to XLIF surgery for their condition will be included. The following eligibility criteria are designed to identify existing clinic patients for whom study under this protocol is considered appropriate. All subjects must meet the inclusion/exclusion criteria below in order to be considered for enrollment.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2014-06; Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Reproducibility of obtaining reliable responses and response thresholds monitored over the course of surgery. | Intraoperative

SECONDARY OUTCOMES:
Correlation of any observed changes in the response or response thresholds with surgical events. | Intraoperative
Correlation between patient characteristics and the ability to generate and reliably record responses and response thresholds. | Intraoperative
Correlation between observed changes in the response or response threshold and postoperative neural status. | 6 weeks postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, MS, Study Director — NuVasive
Locations (2):
- United States (2):
  - Durango Orthopaedics Associates/Spine Colorado, Durango, Colorado
  - Pinnacle Orthopaedics & Sports Medicine Specialists, Marrietta, Georgia

REFERENCES:
- See also: Related Info — http://www.nuvasive.com